CLINICAL TRIAL: NCT06842147
Title: Effectiveness of Artificial IntelliGence-Driven Single-LEad Long-TerM Electrocardiograms MonItoring in Detecting New-Diagnosed Atrial FIbrillation
Acronym: GEMINI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Beijing An Zhen Hospital
Record Dates: First submitted 2025-02-10; First posted 2025-02-24 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; patch
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term Screening Group (Experimental): This group will use the 7-day single-lead ECG monitoring device, a standard 12-lead ECG, family-centered AF education and opportunistic screening.
  Interventions: Device: 7-day single-lead long-term ECG monitoring device.
- Standard Screening Group (Active Comparator): This group will receive a standard 12-lead ECG, family-centered AF education and opportunistic screening.
  Interventions: Device: Standard Screening Group

INTERVENTIONS:
Device: 7-day single-lead long-term ECG monitoring device. — Participants in the long-term screening group will undergo baseline data collection and a 12-lead ECG at baseline, followed using a 7-day single-lead long-term ECG monitoring device. This device continuously collects dynamic ECG data for seven days and allows participants to view and store ECGs through the accompanying software (registration number: 20192070163).
  Arms: Long-term Screening Group
Device: Standard Screening Group — Patients in the standard screening group will undergo baseline data collection and a standard 12-lead ECG at the start of the study, with follow-up including opportunistic ECG checks as needed. Those diagnosed with AF will receive anticoagulation and antiarrhythmic therapy according to clinical guidelines.
  Arms: Standard Screening Group

SUMMARY:
Abstract Purpose: Atrial fibrillation (AF) is a leading cause of stroke and heart failure, yet detection remains suboptimal in rural settings due to limited resources. This study evaluates whether an enhanced screening strategy using artificial intelligence (AI)-integrated 7-day single-lead electrocardiogram (ECG) patches improves AF detection and long-term clinical outcomes compared to routine care in rural China.

Methods: This cluster-randomized trial will be conducted across 128 village clinics in Quzhou, Zhejiang Province. Villages are randomized 1:1 to either enhanced or routine screening. Participants aged 60 years or older (approximately 120 per village) in both arms receive family-centered AF education and opportunistic assessments. The enhanced group undergoes screening via 7-day single-lead ECG patches, while the routine group utilizes standard 12-lead ECGs.

Results: The trial features two primary endpoints. The Phase 1 endpoint is the newly diagnosed AF detection rate during a 1-year screening period. The Phase 2 endpoint is a 3-year composite outcome of all-cause mortality, stroke or systemic embolism, and hospitalization for heart failure.

Conclusion: By integrating wearable AI technology into primary care, this trial seeks to overcome diagnostic barriers in resource-limited environments. The findings will determine if prolonged digital monitoring can significantly enhance AF detection and reduce major cardiovascular events in elderly rural populations.

DETAILED DESCRIPTION:
Effectiveness of Artificial IntelliGence-Driven Single-Lead Long-Term Electrocardiograms Monitoring In Detecting New-Diagnosed Atrial FIbrillation (GEMINI) trial is a parallel, two-stage cluster randomized trial being conducted in 128 villages in Qujiang District, Quzhou City, Zhejiang Province. Village clinics serve as the primary health care units and provide essential services to rural residents, with one clinic allocated to each administrative village in China. Each village clinic is staffed by a village doctor with basic medical training (certificate-level) and operates under the supervision of physicians based at 8 township health centers. These township health centers are, in turn, overseen by a single district-level hospital, forming a three-tier hierarchical healthcare system . This decentralized structure, designed to address the shortage of specialist resources at the village level, enables consistent outreach and sustained medical engagement across rural populations. In this study, the villages (clusters) were randomly assigned to either the enhanced screening group (intervention arm) or the routine screening group (control arm). The coprimary outcomes are the 1-year detection rate of newly diagnosed AF (Phase 1) and a 3-year composite of all-cause mortality, stroke or systemic embolism, and hospitalization for heart failure (Phase 2).

ELIGIBILITY:
Inclusion Criteria:

Age 60 years or older No previous history of atrial fibrillation (AF) Willing to participate in random assignment and follow-up

Exclusion Criteria:

Patients with a pacemaker or implanted cardioverter-defibrillator (ICD) Patients with cognitive impairment or unable to provide informed consent Patients with an estimated life expectancy of less than one year (e.g., advanced cancer or end-stage renal disease) Patients deemed unsuitable for the study by the investigator Patients who refuse to participate

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15360 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Detection rate of new atrial fibrillation diagnoses | 1 year
  Detection rate of new atrial fibrillation diagnoses in both groups. Atrial fibrillation is defined by a single-lead ECG (≥30s) or a 12-lead ECG (≥10s) showing absent P waves, replaced by irregular fibrillation waves (f-waves) of varying size, shape, and duration, and absolute irregularity of RR intervals. Two cardiologists will interpret the ECG, and if there is doubt, a third cardiologist will review the case. Opportunistic ECG is defined as any ECG performed for medical reasons during follow-up (primarily 12-lead ECG), which must be reported and diagnosed.
Composite endpoints | 3 years
  The all-cause mortality, stroke/systemic embolism, and heart failure hospitalization rate in the study population.

SECONDARY OUTCOMES:
Atrial Fibrillation Burden Assessment | 1 year
  Assessment of atrial fibrillation burden, defined by the duration and frequency of episodes, measured through continuous monitoring and ECG evaluations.
All-Cause Mortality Rate | 3 years
  The all-cause mortality rate in the study population, measuring the number of participants who have died from any cause.
Cardiovascular Mortality Rate | 3 years
  The cardiovascular mortality rate, defined as death directly caused by cardiovascular diseases, including acute myocardial infarction, heart failure, stroke, etc.
Stroke/systemic embolism: | 3 years
  Stroke is defined as an acute episode of focal or global neurological dysfunction caused by intraparenchymal, intraventricular, or subarachnoid hemorrhage, or central nervous system infarction. Systemic embolism refers to a thrombus or other material traveling through the bloodstream and causing embolism in other vital organs (e.g., kidneys, limbs, etc.).
Heart Failure Hospitalization Rate | 3 years
  The rate of hospitalization due to heart failure in the study population.
Cardiovascular Hospitalization Rate | 3 years
  The rate of hospitalization due to cardiovascular events (excluding heart failure) in the study population.
Detection Rate of New Atrial Fibrillation | 3 years
  The detection rate of new atrial fibrillation diagnoses during the study period, defined by the criteria set for ECG findings.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Zhejiang, Quzhou, China

IPD SHARING:
Plan to Share IPD: Undecided